CLINICAL TRIAL: NCT07091825
Title: A Prospective, Multi-center, Open-Label, Randomized Controlled, Non-Inferiority Clinical Study Evaluating the Efficacy and Safety of Contact Lens Lubricant in Rigid Gas Permeable Corneal Contact Lens Wearers
Brief Title: Evaluating the Efficacy and Safety of Contact Lens Lubricant in Rigid Gas Permeable Corneal Contact Lens Wearers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Avizor SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Avizor-CT
Record Dates: First submitted 2025-06-26; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tested medical device (Experimental): LACRIFRESH OCU-DRY 0.3% OSD
  Interventions: Device: LACRIFRESH OCU-DRY 0.3% OSD
- Control medical device (Active Comparator): Rigid contact lens lubricant
  Interventions: Device: Rigid contact lens lubricant

INTERVENTIONS:
Device: LACRIFRESH OCU-DRY 0.3% OSD — Use LACRIFRESH OCU-DRY 0.3% OSD as the daily contact lens lubricant product.
  Arms: Tested medical device
Device: Rigid contact lens lubricant — Use Rigid contact lens lubricant as the daily contact lens lubricant product.
  Arms: Control medical device

SUMMARY:
This trial aims to evaluate the safety and effectiveness of LACRIFRESH OCU-DRY 0.3% OSD, a contact lens lubricant produced by AVIZOR, S.A. This clinical trial adopts a Multi-center, randomized, open-label, positive parallel-controlled design in accordance with the principles outlined in the Norms on the Quality Management for the Clinical Trials of Medical Devices issued by the National Medical Products Administration of China.

Meanwhile, following statistical requirements, 152 rigid contact lens wearers are planned to be enrolled after screening and meeting the inclusion criteria. Participants will be randomly assigned to groups and provided with lenses, lubricants, and care solutions accordingly. Clinical follow-up assessments are scheduled at 1 week, 1 month, and 3 months after use.

The primary efficacy indexes are the percentage of patients with binocular comfort score ≥ Level 3 at the 1-month follow-up and the percentage of patients with best corrected distance visual acuity with contact lenses for both eyes ≥5.0 at the 1-month follow-up after using the contact lens lubricant. Secondary efficacy indexes include, best corrected distance visual acuity with lenses, visual acuity with lenses, residual diopter, tear break-up time, uncorrected visual acuity, examination of contact lens fitting status, lens assessment, and contact lens lubricant evaluation during the corresponding follow-up periods. Safety indexes include slit lamp examination, fundus examination, IOP, corneal endothelial cell, adverse events, serious adverse events, device defects that may lead to serious adverse events, other device defects during the corresponding follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 8 and older, no gender limitation;
2. Rigid gas permeable corneal contact lens (OK lens) wearers;
3. The best corrected distance visual acuity of framed lenses in both eyes can reach 5.0 (5-Point Scale);
4. Be able and willing to comply with all treatments and follow-ups;
5. Be able to understand the purpose of the trial, participate voluntarily and have ICF signed by the subject himself/herself or his/her legal guardian.

Exclusion Criteria:

1. Patients with only one eye meeting the inclusion criteria.
2. Patients with abnormal clinical abnormalities or systemic diseases affecting the eyes that occurred or is occurring before screening and, in the investigator's judgment, preclude the use of corneal contact lenses.
3. Patients with some eye diseases that affect contact lens wearing: such as acute or chronic eye diseases, conjunctivitis catarrhalis aestiva, glaucoma, corneal abnormalities, keratoconus, etc.
4. Patients with allergies to the components of contact lens or contact lens care solution involved in this trial;
5. Patients who are using or need to use drugs that may cause dry eyes or affect vision and corneal curvature (e.g. immunosuppressant, glucocorticoids, IOP-lowering drugs, low concentration atropine) during the study;
6. Patients with a history of intraocular operation;
7. Patients with abnormal IOP (the single eye IOP <10 mmHg or >21mmHg, or the IOP difference of both eyes >5mmHg), obvious fundus abnormalities, examination of corneal endothelial cell (abnormal ≥ Level 4), or slit-lamp examination abnormalities.
8. Patients with dry eye syndrome or with break up time (BUT) <5s.
9. Subjects who participated in other drug clinical trials within 90 days before screening, and participated in other medical device clinical trials within 30 days;
10. Patients who wore rigid contact lens (including orthokeratology lens) within the past 30 days;
11. Patients who are pregnant, nursing or planning to conceive at the enrollment;
12. Patients with contraindications for wearing rigid contact lenses or unsuitable for wearing rigid contact lenses as indicated by examination results;
13. Other conditions for which the investigator judged the patient unsuitable for inclusion.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with comfort scores ≥ Level 3 for both eyes at the 1-month follow-up after using the contact lens lubricant. | 1 month
Percentage of subjects with the best corrected distance visual acuity in both eyes with lenses ≥5.0 at the 1-month follow-up after using the contact lens lubricant. | 1 month

SECONDARY OUTCOMES:
Changes in subjective symptoms assessed by subjective acceptability Scale of National Medical Products Administration（NMPA） | 1 week, 1 month, and 3 months
  According to the Guidelines for Registration Review of Contact Lens Care Products of NMPA, subjective acceptability of contact lens care products is investigated through the investigation of subjective symptoms during follow-up, specifically including evaluations of comfort, visual and operability assessments. Higher scores indicate a more favorable outcome for the endpoint. For comfort assessment, the 6-point scale is defined as follows: Level 0: Painful; Level 1: Extremely uncomfortable; Level 2: Mildly uncomfortable; Level 3: Comfortable; Level 4: Very comfortable; Level 5: Excellent. For visual and operability assessments, the 6-point scale is defined as follows: Level 0: Unacceptable; Level 1: Very poor; Level 2: Poor; Level 3: Good; Level 4: Very good; Level 5: Outstanding.
Changes in best corrected distance visual acuity with lenses | 1 week, and 3 months
Changes in lens wearing vision and residual diopter | 1 week, 1 month, and 3 months
Changes in tear break up time (TBUT) | 1 week, 1 month, and 3 months
Changes in uncorrected visual acuity | 1 week, 1 month, and 3 months
Changes in contact lens fitness examination | 1 week, 1 month, and 3 months
Changes in lens assessment | 1 week, 1 month, and 3 months
Changes in contact lens lubricant evaluation | 1 week, 1 month, and 3 months
Changes in slit-lamp examinations | 1 week, 1 month, and 3 months
Changes in fundus examinations | 1 month and 3 months
Comparison between groups for intraocular pressure (IOP) at each follow-up visit, along with changes relative to baseline | 1 week, 1 month, and 3 months
Comparison between groups for examination of corneal endothelial cell at each follow-up visit, along with changes relative to baselineChanges | 3 months
Incidence of adverse events | From the date of randomization until the occurrence of adverse events, assessed for up to 3 months
Incidence of serious adverse event | From the date of randomization until the occurrence of serious adverse event, assessed for up to 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Aier Intech Eye Hospital, Beijing, Beijing Municipality
  - Tianjin Eye Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality